CLINICAL TRIAL: NCT05354687
Title: The Effect of Pressure Injury Assessment Training Given by Self-directed Learning and Small Group Teaching Methods on Nursing Students' Knowledge and Skill Levels
Brief Title: Comparison of Self Directed Learning and Small Group Teaching Methods on Pressure Injury Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sinan Aydoğan, Research Assisstant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: GaziU-SBF-SA-1
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Pressure Ulcer
Keywords: pressure ulcer; self-directed learning; small-group learning; pressure injury; pressure injury assessment
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: a three-group, pre-test - post-test, randomized controlled experimental study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know which group they are in. The knowledge test will be filled online by the participants. A nurse other than the researchers served as an evaluator during the skill assessments. The evaluator is unaware of which group the students belong to. The analysis of the tests data will be done by the statistician. No information will be given to the statistician about which group the participants are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): No intervention will be given to participants. Students will be given pre-test and post-tests.
- Small-group Teaching Group (Experimental): Participants will be given training on the evaluation of pressure injuries with small-group teaching techniques.
  Interventions: Other: Small-group Teaching
- Self-directed Learning Group (Experimental): Participants will be given training on the evaluation of pressure injuries with self-directed learning technique.
  Interventions: Other: Self-directed Learning

INTERVENTIONS:
Other: Small-group Teaching — The Small-group Teaching will include theoretical lectures and laboratory practice. Theoretical training will be given in 2 hours and will last 2 week. After the theoretical training, laboratory practice will be made with mannequins, pressure injury models and photographs in the nursing skills laboratory. Laboratory practices will be done in groups of about 10 students. Laboratory application will take 1 week.
  Arms: Small-group Teaching Group
Other: Self-directed Learning — The training will be given in two stages. The first stage of the training will be given via the mobile application for 2 weeks. Students will be able to access the training individually, wherever and whenever they want, via the mobile application. In the second stage, students will individually conduct laboratory practice. Students who start using the mobile application will make laboratory applications individually, whenever they want when the laboratory is available. Models and materials that students will need will be available in the laboratory. They will be able to get help from the trainer when they need it. Individual laboratory application will take 1 week.
  Arms: Self-directed Learning Group

SUMMARY:
The purpose of this study is to determine the effect of pressure injury assessment training given by self-directed learning and small-group teaching methods on the knowledge and skill levels of nursing students: a three-group, pre-test - post-test, randomized controlled, parallel-group experimental study.

DETAILED DESCRIPTION:
Pressure injury is a common health problem worldwide. The global prevalence of hospital-associated pressure injuries was 8.4%. Regular wound assessment is required to determine appropriate treatment methods, monitor wound healing, and identify complications early in the pressure injury treatment process in order to achieve clinical goals.

According to the literature, nurses and nursing students have a low level of knowledge about pressure injury and there is a knowledge gap between nurses' knowledge of pressure injury and pressure injury practices. As a result, it is necessary to teach skills so that they can put their knowledge into practice. Individuals born after 2000, referred to as Generation Z, make up the majority of students beginning undergraduate education today. The most significant difference between Generation Z and other generations is that they were born during a period when digital high technology was widely used. This generation, also known as the "Internet generation," is constantly surrounded by new technological opportunities, communication, and transportation facilities. Because of these characteristics, it is critical to use teaching methods that will appeal to them when educating students in this group.

In a classroom, there are fast and slow learners. The amount of time allotted to students naturally decreases as the number of students in the class grows. Furthermore, student differences prevent the entire class from learning at the same time. Some students do not learn right away, others later, and still others do not learn at all in such a classroom. Education should be personalized in order to eliminate all of these non-occurrences.With the widespread use of smart phones today, mobile learning has become commonplace. Students gain clinical practice skills and experience when mobile technology is used as a support tool in nursing education practices.

For this purpose, the trainings to be given with the mobile application in this study will be supported by the activities in which the students can practice individually in the skill laboratory.

ELIGIBILITY:
Inclusion Criteria:

* To be registered for the Nursing Vocational Application Course
* Volunteering to participate in the research
* Having a mobile device (smartphone, tablet PC etc.)

Exclusion Criteria:

* To have received training on the evaluation of pressure injuries other than the basic nursing education

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of Pressure Injuries Knowledge Test | five weeks
  The knowledge test was developed by the researchers in line with the literature. Learning objectives on the assessment of pressure injuries were determined and a table of specifications was prepared. A total of 34 questions were prepared, with at least 3 questions for each learning objective. For the knowledge test created, expert opinions were obtained from 6 faculty members in the field of nursing principles and 3 certified ostomy and wound care nurses. Within the scope of the research, the knowledge test will be applied to at least 100 3rd year nursing students and the item difficulty and discrimination indexes will be examined. If necessary, questions will be revised or removed from the test.
Pressure Injury Evaluation Form | five weeks
  The pressure injury evaluation form was developed by researchers based on the "Wound diagnosis evaluation and follow-up form" of the Wound Ostomy Incontinence Nurses Association and pressure injury staging form developed by National Pressure Injury Advisory Panel (NPIAP). The form, which includes the staging and evaluation of pressure injury, consists of the subheadings of the wound bed and the wound periphery. The expert opinion of the form was obtained from three faculty members who are experts in the Department of Nursing Fundamentals and two specialist nurses who are actively working as wound care nurses, who have a Stoma and Wound Care Certificate approved by the Ministry of Health. This form will be used in the assessment of pressure injuries skills assessment.

SECONDARY OUTCOMES:
Pressure Injuries Assessment Education Evaluation Form | 1 week
  In this form, students express their opinions about the Evaluation of Pressure Injuries training and mobile application. The section on the Evaluation of Pressure Injuries training consists of open-ended questions. The other section is a 5-point Likert-type section with 19 statements about the mobile application. Positive statements are items 1, 3, 5, 6, 8, 10, 11, 13, 14, 16, 17, and 19, while negative statements are items 2, 4, 7, 9, 12, 15, and 18. Each item on the form is scored separately. Each item is worth a minimum of one point and a maximum of five points. Higher scores for positive items mean better outcome, and higher scores for negative items mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nurcan Çalışkan, Professor, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sezgünsay, E. Hemşirelik öğrencilerinin basınç yaralanması değerlendirme becerilerinin geliştirilmesinde yüksek gerçeklikli simülasyon yönteminin etkinliğinin incelenmesi, 2019 (Master's thesis, Gülhane Sağlık Bilimleri Enstitüsü).
- [Derived] Aydogan S, Caliskan N. The effect of self-directed learning via a smartphone application and small-group teaching on nursing students' learning of pressure injury assessment: A randomized controlled study. Nurse Educ Pract. 2025 May;85:104336. doi: 10.1016/j.nepr.2025.104336. Epub 2025 Mar 27. PMID 40187051